CLINICAL TRIAL: NCT00703300
Title: Phase I Study of Decitabine (Dacogen) and Bortezomib (Velcade) in Acute Myeloid Leukemia
Brief Title: Decitabine and Bortezomib in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00263; NCI-2009-00263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-08047; 2008C0034; CDR0000598089; 08047 (Other: Ohio State University Medical Center); 8008 (Other: CTEP); U01CA076576 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Bortezomib; Decitabine

ARMS (1):
- Treatment (enzyme inhibitor therapy and chemotherapy) (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 or 1-10 and bortezomib IV on days 5 and 8 or days 5, 8, 12, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Once the maximum tolerated dose is determined, an additional 6 patients are treated at the recommended phase II dose.
  Interventions: Drug: bortezomib; Drug: decitabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of bortezomib when given together with decitabine in treating patients with acute myeloid leukemia. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with decitabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of bortezomib (Velcade, PS-341) in combination with decitabine in patients with acute myeloid leukemia (AML) II. To define the specific toxicities and the dose limiting toxicity (DLT) of decitabine plus bortezomib combination

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR). II. To determine the rate of complete remission (CR) of decitabine plus bortezomib in AML III. To correlate the biological activity of decitabine as demethylating agent (changes in target gene methylation and gene expression, DNMT1 protein expression, global methylation) with clinical endpoints and plasma pharmacokinetics of decitabine.

IV. To characterize the biological activity of bortezomib as a potential demethylating agent V. To correlate intracellular concentration of decitabine-triphosphate with global DNA methylation and other biological endpoints as well as clinical response.

VI. To explore the biologic role of microRNAs in determining clinical response to the decitabine plus bortezomib combination and achievement of the other pharmacodynamic endpoints.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive decitabine intravenously (IV) over 1 hour on days 1-5 or 1-10 and bortezomib IV on days 5 and 8 or days 5, 8, 12, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Once the maximum tolerated dose is determined, an additional 6 patients are treated at the recommended phase II dose.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML), meeting one of the following criteria:

  * Relapsed or refractory disease (≥ 18 years of age)
  * Previously untreated disease (≥ 60 years of age)
* Secondary AML or therapy-related AML allowed
* No granulocytic sarcoma as the sole site of disease
* No active or relapsed CNS disease
* No advanced malignant solid tumors
* ECOG performance status 0-2
* Life expectancy > 6 months (if patient has co-morbid illness)
* Total bilirubin < 2.0 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with HIV infection are eligible provided the following criteria are met:

  * No history of AIDS
  * Has a sufficiently high CD4 count (> 400/mm³)
  * Has low HIV viral loads (< 30,000 copies/mL plasma)
  * Does not require anti-HIV therapy
* No uncontrolled active infection
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to decitabine or bortezomib that are not easily managed
* No hypersensitivity to boron or mannitol
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable or uncontrolled angina pectoris
  * Serious cardiac arrhythmia
  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Severe uncontrolled ventricular arrhythmias
  * Acute ischemia or active conduction system abnormalities by ECG
* No serious medical or psychiatric illness or social situation that would preclude participation in this study
* No pre-existing neuropathy ≥ grade 2
* No other serious neurologic toxicity that would significantly increase the risk of complications from bortezomib therapy
* Recovered from prior therapy (toxicity < grade 2)
* More than 14 days since prior investigational agents
* More than 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy
* Prior decitabine or azacitidine for myelodysplastic syndromes (MDS) or AML allowed
* More than 6 months since prior decitabine, azacitidine, or bortezomib
* No concurrent palliative radiotherapy
* No other concurrent investigational agents
* No other concurrent direct anti-leukemia therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of bortezomib in combination with decitabine | During course 1 (28 days)
  If a patient meets the definition of dose-limiting toxicity (DLT), the patient may continue on with study therapy provided that the toxicity can be managed according to the dose modification guidelines. For DLT = 2, dose level will stop. This dose level will be declared the MTD administered dose (highest dose administered). As an exploratory, phase I study, no inferential statistical tests of hypotheses are planned. Data collected will be descriptive and provide limited estimates of variability given the small sample sizes at each dose level.
Specific toxicities | Up to 30 days post-treatment
  Toxicity will be characterized using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. As an exploratory, phase I study, no inferential statistical tests of hypotheses are planned. Data collected will be descriptive and provide limited estimates of variability given the small sample sizes at each dose level.
DLT of bortezomib in combination with decitabine | During course 1 (28 days)
  Toxicity will be characterized using the National Cancer Institute CTCAE version 3.0. As an exploratory, phase I study, no inferential statistical tests of hypotheses are planned. Data collected will be descriptive and provide limited estimates of variability given the small sample sizes at each dose level.

SECONDARY OUTCOMES:
Overall response rate | Up to 30 days post-treatment
  Assessment of clinical response will be made according to International Working Group criteria. The major criteria for judging response will include physical examination and examination of blood and bone marrow.
Rate of complete remission (CR) | Up to 30 days post-treatment
  The major criteria for judging response will include physical examination and examination of blood and bone marrow (morphologic CR and cytogenetic CR)

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Blum W, Schwind S, Tarighat SS, Geyer S, Eisfeld AK, Whitman S, Walker A, Klisovic R, Byrd JC, Santhanam R, Wang H, Curfman JP, Devine SM, Jacob S, Garr C, Kefauver C, Perrotti D, Chan KK, Bloomfield CD, Caligiuri MA, Grever MR, Garzon R, Marcucci G. Clinical and pharmacodynamic activity of bortezomib and decitabine in acute myeloid leukemia. Blood. 2012 Jun 21;119(25):6025-31. doi: 10.1182/blood-2012-03-413898. Epub 2012 May 7. PMID 22566605